CLINICAL TRIAL: NCT03951142
Title: Imaging Perfusion Restrictions From Extracellular Solid Stress - An Open-label Losartan Study
Acronym: ImPRESS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kyrre Eeg Emblem (Other)
Responsible Party: Sponsor-Investigator, Kyrre Eeg Emblem, Coordinating investigator, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ImPRESS; 2018-003229-27 (EudraCT Number)
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Glioblastoma; Brain Metastases
Keywords: Magnetic Resonance Imaging; Brain Cancer; Angiotensin II receptor blocker; Losartan; Perfusion; Solid stress
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: An open-label, single institutional phase II trial with an individual stepped-wedge, randomized, assessor-blinded, dose-finding design on three indications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study A: Recurrent glioblastoma (denoted 'AR') (Experimental): Patients with recurrent glioblastoma (N=54) with be randomized (ratio 1:1:1) to doses of 25mg, 50mg or 100mg daily of losartan while on treatment. Losartan (tablet) will be administered every day, with 2 weeks (14 consecutive days) defined as a treatment cycle. Based on randomization, a minimum of three cycles and a maximum of 12 cycles will be administered for a total of 6 weeks (42 days) to 24 weeks (168 days), respectively. Patients randomized to 100mg of losartan will all receive treatment for the maximum duration.
  A stepped-wedge randomized design (ratio 1:1:1 for all doses over the three first cycles) is proposed to compare participants on- and off- study IMP and assess any dose-response relationship losartan. This study arm will also investigate any additional long-term beneficial effects of losartan while receiving chemotherapy (temozolomide or lomustine tablets).
  Interventions: Drug: Losartan
- Study A: Newly diagnosed glioblastoma (denoted 'AN') (Experimental): Patients with newly diagnosed glioblastoma (N=54) with be randomized (ratio 1:1:1) to doses of 25mg, 50mg or 100mg daily of losartan while on treatment. Losartan (tablet) will be administered every day, with 2 weeks (14 consecutive days) defined as a treatment cycle. Based on randomization, a minimum of three cycles and a maximum of 17 cycles will be administered for a total of 6 weeks (42 days) to 34 weeks (238 days), respectively. Patients randomized to 100mg of losartan will all receive treatment for the maximum duration.
  A stepped-wedge randomized design (ratio 1:1:1 for all doses over the three first cycles) is proposed to compare participants on- and off- study IMP and assess any dose-response relationship losartan. This study arm will also investigate any additional long-term beneficial effects of losartan while receiving adjuvant chemotherapy (Temozolomide tablets).
  Interventions: Drug: Losartan
- Study B: Brain metastases (denoted 'BM') (Experimental): Patients with brain cancer from non-small cell lung cancer (N=45) with all receive a dose of 50mg daily of losartan while on treatment. Losartan (tablet) will be administered every day, with 3 months (90 consecutive days) defined as a treatment cycle. A minimum of one cycle and a maximum of three cycles will be administered for a total of 3 months (90 days) to 9 months (270 days), respectively.
  A stepped-wedge randomized design (ratio 1:1:1 over the three first cycles) is proposed to compare participants on- and off- study IMP and assess any dose-response relationship losartan. This study arm will also investigate any additional long-term beneficial effects of losartan while receiving chemotherapy alone (carboplatin in combination with vinorelbin or pemetrexed or equivalent analogs) or in combination with pembrolizumab (2mg/kg/3rd week).
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — This trial is open-label; therefore, the participant, the trial site personnel, the Sponsor and/or designee are not blinded to treatment. Drug identity (name, strength) is included in the label text. Storage, handling and preparation requirements will be handled in concordance with the Pharmacy Manual for losartan.

SUMMARY:
An open-label, single institutional phase II trial of losartan in patients with primary and metastatic brain tumors with an individual stepped-wedge, randomized, assessor-blinded, dose-finding design on three indications.

DETAILED DESCRIPTION:
For this study losartan, an angiotensin-II inhibitor, is defined as the Investigational Medicinal Product (IMP). The focus of the study is to assess the dose-response relationship of losartan on imaging-based measures of tissue perfusion and mechanical forces in patients with brain tumors. We hypothesize that losartan improves the effect of traditional cancer treatment by alleviating mechanical forces (solid stress) of the tumor microenvironment to improve tissue perfusion, while administration of losartan alone has little effect on cancer patients.

This is an open-label study and no active comparator or placebo will be used. Study participants include adult patients with newly diagnosed- and recurrent glioblastoma, as well as adult patients with metastatic brain tumors from non-small cell lung cancer. The study will assess the safety of losartan treatment and its dose-response relationship on conventional and experimental radiographic characteristics when used alone or as an add-on to standard cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically confirmed intracranial glioblastoma, WHO grade 4 (Study A), or a minimum of one radiographically confirmed metastasis to the brain from a primary non-small-cell lung cancer (Study B)
2. Ability to undergo an MRI exam, including administration of a standard clinical dose of an MRI-specific contrast agent of gadolinium or similar
3. Measurable intracranial disease (Study A - recurrent glioblastoma, and Study B only), defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm with MRI
4. Age ≥18 years
5. Eligible for administration of the active substance (losartan) in concordance with study protocol, the criteria of the product label (Cozaar) and deemed fit for trial by the treating physician.
6. An ECOG performance status of ≤2 or equivalent KPS of ≥60%
7. Life expectancy from start of treatment of more than 3 months
8. Previous history of neurosurgical procedure (Study A - only) or stereotactic radiosurgery and immunotherapy (Study B) at time of study inclusion
9. Scheduled for chemotherapy and/or radiotherapy and/or stereotactic radiosurgery (Study A - recurrent glioblastoma), neurosurgery, radiotherapy and chemotherapy (Study A - newly diagnosed glioblastoma), immunotherapy and/or chemotherapy (Study B)
10. Pre-study documentation on O6-methylguanin-DNA-methyltransferase (MGMT) promoter methylation status and on the isocitrate dehydrogenase (IDH) gene mutation status of their disease (study A only)
11. Organ functions of sufficient quality and robustness to undergo study treatment as determined by the study principal investigator (PI) or designee
12. Female patients of childbearing potential (postmenarcheal, not postmenopausal (>12 continuous months of amenorrhea with no identified cause other than menopause), and no surgical sterilization) should use highly effective contraception and take active measures to avoid pregnancy while undergoing IMP treatment and for at least 14 days after the last dose. Birth control methods considered to be highly effective include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence when it is the preferred and usual lifestyle of the subject.
13. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Hypersensitivity to the active substance (losartan) or to any of the excipients
2. Patients on antihypertensive agents that cannot be substituted with losartan.
3. Patients on medication that may induce hypotension and/or increase potassium levels and/or cause metabolism-related pharmacokinetic drug-drug interactions with losartan. If medication with such effects can safely be discontinued or replaced, the patient can be included in the study after a washout period before baseline.
4. Patients with hepatic or renal impairment of any reason
5. Patients with symptomatic hypotension of any reason
6. Patients with primary hyperaldosteronism
7. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption should not take this medicine
8. Inadequate recovery from toxicity and/or complications of previous therapy as determined by the treating physician
9. Patients with evidence of recurrence inside the radiotherapy target volume less than 3 months since last radiotherapy fraction (Study A - recurrent glioblastoma only)
10. For Study B subjects only. A diagnosis of immunodeficiency or hypersensitivity to the PD-1 inhibitors or any of its excipients
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, coronary heart disease and cerebrovascular disease, unstable angina pectoris, cardiac arrhythmia, angioedema, intravascular volume depletion, or psychiatric illness/social situations that would limit compliance with study requirements as determined by treating the physician
12. Patients suffering from aortic or mitral stenosis, or obstructive hypertrophic cardiomyopathy
13. Patient with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study as determined by the treating physician
14. Pregnant or breastfeeding patient
15. Known additional active non-study related malignancy
16. Applies to Study B patients qualifying for immunotherapy only: Active autoimmune disease that has required systemic treatment in the last 2 years (including use of non-study related disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed
17. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
18. Unable to undergo brain MRI according to study protocol
19. For Study B subjects only: No previous history of immunotherapy at time of study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative cerebral blood flow by MRI | Study AR: Baseline, Day 14-16, Day 28-30, Day 42-44. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44. Study arm BM: Baseline, Day 90±7, Day 180±7, Day 270±7
  Change from baseline in the radiographic biomarker relative cerebral blood flow (rCBF)
Relative solid stress by MRI | Study AR: Baseline, Day 14-16, Day 28-30, Day 42-44. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44. Study arm BM: Baseline, Day 90±7, Day 180±7, Day 270±7
  Change from baseline in the radiographic biomarker relative solid stress

SECONDARY OUTCOMES:
Relative cerebral blood volume by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative cerebral blood volume (rCBV)
Mean transit time by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative mean transit time (rMTT)
Contrast agent extravasation by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker contrast agent extravasation
Relative vessel size index by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative vessel size index
Relative mean vessel density by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative mean vessel density
Relative mean vessel caliber by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative mean vessel caliber
Apparent diffusion coefficient by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker apparent diffusion coefficient
Fractional anisotropy by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker fractional anisotropy
Relative shear modulus by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative shear modulus
Relative stiffness by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative stiffness
Relative viscosity by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative viscosity
Relative strain tensor by MRI | Study arm AR: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 78-8/+1, Day 162-8/+1. Study arm AN: Baseline, Day 14-16, Day 28-30, Day 42-44, Day 148-8/+1, Day 232-8/+1. Study arm BM: Baseline, Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in the radiographic biomarker relative strain tensor
Drug tolerance | Study arm AR: Day 168+14. Study arm AN: Day 238+14. Study arm BM: Day 270+14.
  Drug tolerance of losartan according to NCI-CTCAE v4.0
Neurologic performance by KPS | Study arm AR: Baseline, Day 14-16, Day 42-44, Day 85±4, Day 169±4. Study arm AN: Baseline, Day 14-16, Day 42-44, DAy 71±4, Day 155±4, Day 239±. Study arm BM: Baseline, Day 90-7, Day 180-1, Day 270-1, Day 360±7
  Change from baseline in neurologic performance scores by Karnofsky Performance Score (KPS). Range from [00-0]. The lower the Karnofsky score, the worse the survival for most serious illnesses.
Neurologic performance by ECOG | Study arm AR: Baseline, Day 14-16, Day 42-44, Day 85±4, Day 169±4. Study arm AN: Baseline, Day 14-16, Day 42-44, DAy 71±4, Day 155±4, Day 239±. Study arm BM: Baseline, Day 90-7, Day 180-1, Day 270-1, Day 360±7
  Change from baseline in neurologic performance scores by Eastern Cooperative Oncology Group (ECOG) scores. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability in a range from 0 (best) to 5 (dead).
Neurologic performance by NANO | Study arm AR: Baseline, Day 14-16, Day 42-44, Day 85±4, Day 169±4. Study arm AN: Baseline, Day 14-16, Day 42-44, DAy 71±4, Day 155±4, Day 239±. Study arm BM: Baseline, Day 90-7, Day 180-1, Day 270-1, Day 360±7
  Change from baseline in neurologic performance scores by Neurologic Assessment in Neuro-Oncology (NANO) scale as an objective and quantifiable metric of neurologic function evaluable during a routine office examination. The NANO Scale evaluates 9 major domains of neurologic function, with each domain being scored on a range from 0 to 2 or 3.
RANO | Study arm AR: Day 78-8/+1, Day 162-8/+1. Study arm AN: Day 148-8/+1, Day 232-8/+1. Study arm BM: Day 90±14, Day 180±14, Day 270±14.
  Change from baseline in radiographic status on MRIs of intracranial disease corresponding to treatment response using the Response Assessment in Neuro-Oncology (RANO) criteria.
Steroid dosage | Study arm AR: Baseline, Days 1-3, 29-31, 57±7, 85±7, 113±7, 141±7, 169±7. Study arm AN: Baseline, Days 29-31, 43-45, 71±7, 99±7, 127±7, 155±7, 183±7, 211±7, 239±7. Study arm BM: Baseline, Days 90±7, 180±7, 270±7, 360±7.
  Change in dosage during study treatment.
Quality of life (QoL) | Study arm AR: Baseline, Day 42-44, 169±4. Study arm AN: Baseline, Day 42-44, Day 155±4, Day 239±4. Study arm BM: Baseline, Day 90-7, Day 180-7, Day 270-7, Day 360±7
  Change from baseline in the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ BN20). It scores 20 items that assess future uncertainty, visual disorder, motor dysfunction, and communication deficit. Items are presented as questions on a scale ranging from 1 = "not at all" to 4 = "very much."
Progression free survival (PFS) | All studies: Day +180, up to 24 months
  6-months progression free survival (6M-PFS) and within 2 years
Overall survival (OS) | All studies: at 12 months, at 24 months, up to 24 months.
  12-months overall survival (12M-OS), 24-months overall survival (24M-OS) and within 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Petter Brandal, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) will be made available at the time of research data publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Supporting information will be made available at the time of research data publication. No end date for sharing of supporting information.
Access Criteria: Open upon request or by journal criteria

REFERENCES:
- [Derived] Lysvik EK, Mikalsen LTG, Rootwelt-Revheim ME, Emblem KE, Hjornevik T. Optimization of Q.Clear reconstruction for dynamic 18F PET imaging. EJNMMI Phys. 2023 Oct 20;10(1):65. doi: 10.1186/s40658-023-00584-1. PMID 37861929